CLINICAL TRIAL: NCT06851611
Title: An Open Short-term Clinical Pilot Trial on Safety and Immunogenicity of Nasal COVID-19 Vaccine at Different Dose Levels and Administration Methods
Brief Title: The Safety and Antibody Response of the Nasal COV2 Vaccine Against the SARS-CoV-2 Virus
Acronym: COV2NOSE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rokote Laboratories Finland Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: COV2FIN11; 2023-509725-49-00 (EU CTIS Number); U1111-1299-1228 (Other: World Health Organization; Universal Trial Number (UTN))
Record Dates: First submitted 2025-02-24; First posted 2025-02-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: COVID19, Sars-Cov-2
Keywords: nasal vaccine; adeno-vectored vaccine; mucosal vaccine; Sars-CoV-2; COVID19
MeSH Terms: conditions — COVID-19 | interventions — COVID-19 Vaccines; Floors and Floorcoverings; Nasal Sprays

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Booster - COV2 Low Dose Level - Nasal Drops (Experimental): Subjects with prior vaccination with at least two doses of any COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccine, low dose level; Other: Nasal Drops
- Booster - COV2 Low Dose Level - Nasal Spray (Experimental): Subjects with prior vaccination with at least two doses of any COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccine, low dose level; Other: Nasal Spray
- Booster - COV2 High Dose Level - Nasal Drops (Experimental): Subjects with prior vaccination with at least two doses of any COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccine, high dose level; Other: Nasal Drops
- Booster - COV2 High Dose Level - Nasal Spray (Experimental): Subjects with prior vaccination with at least two doses of any COVID-19 vaccine
  Interventions: Biological: COVID-19 vaccine, high dose level; Other: Nasal Spray
- Prime - COV2 High Dose Level - Nasal Drops (Experimental): Subjects with no prior COVID-19 vaccination - COULD NOT BE RECRUITED
  Interventions: Biological: COVID-19 vaccine, high dose level; Other: Nasal Drops
- Prime - COV2 High Dose Level - Nasal Spray (Experimental): Subjects with no prior COVID-19 vaccination - COULD NOT BE RECRUITED
  Interventions: Biological: COVID-19 vaccine, high dose level; Other: Nasal Spray

INTERVENTIONS:
Biological: COVID-19 vaccine, low dose level — Test article
  Other Names: COV2
  Arms: Booster - COV2 Low Dose Level - Nasal Drops; Booster - COV2 Low Dose Level - Nasal Spray
Biological: COVID-19 vaccine, high dose level — Test article
  Other Names: COV2
  Arms: Booster - COV2 High Dose Level - Nasal Drops; Booster - COV2 High Dose Level - Nasal Spray; Prime - COV2 High Dose Level - Nasal Drops; Prime - COV2 High Dose Level - Nasal Spray
Other: Nasal Drops — Method of administration of test article
  Arms: Booster - COV2 High Dose Level - Nasal Drops; Booster - COV2 Low Dose Level - Nasal Drops; Prime - COV2 High Dose Level - Nasal Drops
Other: Nasal Spray — Method of administration of test article
  Arms: Booster - COV2 High Dose Level - Nasal Spray; Booster - COV2 Low Dose Level - Nasal Spray; Prime - COV2 High Dose Level - Nasal Spray

SUMMARY:
COV2 is a nasal, investigational vaccine against COVID-19, based on a serotype 5 adenoviral vector producing the SARS-CoV-2 spike protein. In this trial, the primary comparison in terms of safety and immunogenicity will be between two different dose levels of COV2 booster vaccine (low, high), and two different administration methods (nasal drops, nasal spray). In addition, COV2 vaccine will also be evaluated in vaccine naive subjects.

ELIGIBILITY:
Inclusion Criteria

1. Has voluntarily signed the written informed consent
2. 18-75 years old
3. Good general health
4. a) Prior vaccination with at least two doses of any COVID-19 vaccine, OR b) No prior COVID-19 vaccination

Exclusion Criteria

1. Pregnant, planning to become pregnant or breastfeeding women
2. COVID-19 infection within the last nine (9) months
3. Any other vaccination within the last two (2) months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2025-01-21 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-06-26 (Actual)

PRIMARY OUTCOMES:
Primary Immunogenicity | 28 days from baseline
  Percentage of subjects demonstrating a rise in SARS-CoV-2 serum NAb titers against Omicron BA.5 variant
Primary Safety | 28 days from baseline
  Treatment-emergent expected and unexpected adverse effects

SECONDARY OUTCOMES:
Secondary Immunogenicity | 28 days from baseline
  Percentage of subjects demonstrating a rise in SARS-CoV-2 serum NAb titers against Wuhan and JN.1 variants

CONTACTS AND LOCATIONS:
Overall Officials: Seppo Ylä-Herttuala, MD, PhD, Study Director — Rokote Laboratories Finland Oy; Erkko Ylösmäki, PhD, Study Director — Rokote Laboratories Finland Oy
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No